CLINICAL TRIAL: NCT00135486
Title: Evaluate Immunogenicity, Reactogenicity, Safety of GSK Biologicals' MenC-TT Vaccine (2 Formulations) Given With Infanrix Hexa® + GSK Biologicals' Hib MenC-TT Vaccine (2 Formulations) Given With Infanrix Penta® to Infants in Mths 3,4,5 of Life
Brief Title: Study to Evaluate GlaxoSmithKline (GSK) Biologicals' MenC-TT Vaccine and Hib-MenC-TT Vaccine in Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 711202/001
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Infections, Meningococcal
Keywords: Haemophilus Influenzae type b/Meningococcal vaccine; Prophylaxis meningococcal serogroup C disease, Hib diseases
MeSH Terms: conditions — Meningococcal Infections

INTERVENTIONS:
Biological: MenC-TT
Biological: Hib-MenC-TT
  Other Names: MenC-TT

SUMMARY:
The purpose of this primary vaccination study is to evaluate the immunogenicity, safety and reactogenicity of three doses of GSK Biologicals' MenC-TT (Neisseria meningitidis group C polysaccharide-tetanus toxoid) vaccine (2 different formulations) and of three doses of GSK Biologicals' Hib-MenC-TT (Haemophilus influenzae type b-MenC-TT) vaccine (2 different formulations) when given to infants in their 3rd, 4th, and 5th months of life. Concomitant vaccines were given to all children to complete the vaccination agenda.

DETAILED DESCRIPTION:
Five parallel treatment groups receiving a 3-dose primary vaccination course: MenC-TT vaccine (2 formulations, double-blind) + Infanrix hexa® OR Hib-MenC-TT (2 formulations double-blind) + Infanrix penta® OR Meningitec™ + Infanrix hexa® (control). Three blood samples taken, before dose 1 and one month after dose 2 and dose 3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female infants, 8 to 16 weeks of age at the time of the first vaccination.

Exclusion Criteria:

* Previous vaccination against OR history of OR exposure since birth to diphtheria, pertussis, tetanus, polio, hepatitis B, Hib and/or meningococcal disease.
* Planned administration/administration of a vaccine not foreseen in the study since birth.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of any neurologic disorders or seizures, allergic disease or reactions likely to be exacerbated by any component of the vaccine

Ages: 8 Weeks to 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2002-03; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of Meningococcal C serum bactericidal assay using rabbit complement (rSBA-MenC) antibody titers ≥ 1:8 & ≥ 1:128 and titers | Prior to vaccination, one month after the 2nd and 3rd vaccine doses
Evaluation of anti-polysaccharide C (anti-PSC) antibody concentrations ≥ 0.3 µg/mL & ≥ 2 µg/mL and concentrations | Prior to vaccination, one month after the 2nd and 3rd vaccine doses
Evaluation of anti-polyribosyl ribitol phosphate (anti-PRP) antibody concentrations ≥ 0.15 µg/mL & ≥ 1 µg/mL and concentrations | Prior to vaccination, one month after the 2nd and 3rd vaccine doses
Evaluation of anti-diphtheria antibody concentrations ≥ 0.1 IU/mL by ELISA | Prior to and one month after the 3rd vaccine dose
Evaluation of anti-tetanus antibody concentrations ≥ 0.1 IU/mL | Prior to and one month after the 3rd vaccine dose
Evaluation of anti-hepatitis B surface antigen (anti-HBs) antibody concentrations ≥ 10 mIU/mL | Prior to and one month after the 3rd vaccine dose
Evaluation of anti-poliovirus types 1, 2 and 3 antibody titers ≥ 8 mIU/mL | Prior to and one month after the 3rd vaccine dose
Vaccine response to pertussis toxoid (PT) | Prior to 3rd vaccine dose
Evaluation of anti-diphtheria antibody concentrations | Prior to 3rd vaccine dose
Anti-poliovirus types 1, 2 and 3 antibody titers | Prior to and one month after the 3rd vaccine dose
Occurrence of solicited local injection site symptoms | During the solicited follow-up period (Day 0 7) following administration of each vaccine dose
Occurrence of solicited systemic symptoms | During the solicited follow-up period (Day 0 7) following administration of each vaccine dose
Occurrence of unsolicited non-serious adverse events (AEs) | Within one month (Day 0 30) after each vaccination
Occurrence of any serious adverse events (SAEs) | Throughout the entire study period up to and including one month (maximum 30 days) after the last vaccine dose
Vaccine response to pertussis toxoid (PT) | One month after the 3rd vaccine dose
Vaccine response to filamentous haemagglutinin (FHA) | Prior to 3rd vaccine dose
Vaccine response to filamentous haemagglutinin (FHA) | One month after the 3rd vaccine dose
Vaccine response to pertactin (PRN) | Prior to 3rd vaccine dose
Vaccine response to pertactin (PRN) | One month after the 3rd vaccine dose
Evaluation of anti-diphtheria antibody concentrations | One month after the 3rd vaccine dose
Evaluation of anti-tetanus antibody concentrations | Prior to 3rd vaccine dose
Evaluation of anti-tetanus antibody concentrations | One month after the 3rd vaccine dose
Evaluation of anti-HBs antibody concentrations | Prior to 3rd vaccine dose
Evaluation of anti-HBs antibody concentrations | One month after the 3rd vaccine dose
Evaluation of anti-PT antibody concentrations | Prior to 3rd vaccine dose
Evaluation of anti-PT antibody concentrations | One month after the 3rd vaccine dose
Evaluation of anti-FHA antibody concentrations | Prior to 3rd vaccine dose
Evaluation of anti-FHA antibody concentrations | One month after the 3rd vaccine dose
Evaluation of anti-PRN antibody concentrations | Prior to 3rd vaccine dose
Evaluation of anti-PRN antibody concentrations | One month after the 3rd vaccine dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Schmitt HJ, Maechler G, Habermehl P, Knuf M, Saenger R, Begg N, Boutriau D. Immunogenicity, reactogenicity, and immune memory after primary vaccination with a novel Haemophilus influenzae-Neisseria meningitidis serogroup C conjugate vaccine. Clin Vaccine Immunol. 2007 Apr;14(4):426-34. doi: 10.1128/CVI.00377-06. Epub 2007 Feb 7. PMID 17287313
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 711202/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 711202/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 711202/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 711202/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 711202/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 711202/001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register